CLINICAL TRIAL: NCT06514001
Title: A Phase 2, Open Label, Study of AMDX-2011P as a Retinal Tracer in Participants With Alzheimer's Disease
Brief Title: A Study of AMDX-2011P in Participants With Alzheimer's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amydis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMDX-2011P-204
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
Keywords: AD
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMDX-2011P 100 milligram (Experimental): AMDX2011P 100 milligram (4 milliliter) single bolus injection intravenous for diagnostic review
  Interventions: Drug: AMDX-2011P

INTERVENTIONS:
Drug: AMDX-2011P — AMDX-2011P single bolus injection intravenous for diagnostic review

SUMMARY:
The purpose of this study is to assess safety, tolerability, plasma pharmacokinetics and biologic activity of a single intravenous dose of AMDX-2011P in participants with Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
This open-label, masked endpoint assessment study will evaluate the safety, tolerability, plasma pharmacokinetics (PK) and biological activity of an intravenous (IV) dose of AMDX-2011P in participants with AD. Assessments of retinal images will be conducted by central masked assessors.

Participants will be admitted to the study site where eye examination and retinal imaging will be conducted before administration of the study drug. AMDX-2011P will be administered through a single IV bolus injection followed by safety assessments, retinal imaging and PK blood collection.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Alzheimer's Disease (AD) with documented positive amyloid beta signal via positron emission tomography (PET) brain scan
2. Must be willing to consent to genotyping for apolipoprotein E (APOE)
3. Ability to fixate and undergo retinal imaging of both eyes

Exclusion Criteria:

1. Presence of any underlying physical or psychological medical condition that, in the opinion of the investigator, would make it unlikely that the participant will complete the study per protocol
2. Diagnosis of glaucoma, or suspect of having glaucoma in either eye as determined by an ophthalmologist as a clinical investigator, based on results from the eye examination, visual field, and/or optical coherence tomography (OCT) results
3. Diagnosis of intermediate dry, wet/neovascular, or geographic atrophy forms of age-related macular degeneration (AMD) in either eye, OR as determined by an ophthalmologist as a clinical investigator, based on results from the eye examination and/or optical coherence tomography (OCT) results
4. Clinically significant laboratory abnormalities as assessed by the investigator
5. Prolonged QTcF (corrected QT interval by Fridericia method) (>450 ms for males and >470 ms for females), cardiac arrhythmia, or any clinically significant abnormality in the resting electrocardiogram (ECG), as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
AMDX-2011P Adverse Events Profile | 8 days
  Incidence, nature and severity of adverse events/serious adverse events (AEs/SAEs)

SECONDARY OUTCOMES:
Concentration of AMDX-2011P | 2 hours
  Plasma Pharmacokinetic (PK) Concentration (CMax) AMDX-2011P to AMDX-2011
Pharmacokinetic Analysis of AMDX-2011P | 2 hours
  Area under the plasma versus time curve (AUC)
Biological Activity | 8 days
  Detection of amyloid deposits in the retina after intravenous AMDX-2011P administration

CONTACTS AND LOCATIONS:
Overall Officials: David Bingaman, DVM, PhD, Study Director — Amydis Inc.
Locations (3):
- United States (3):
  - Associated Retina Consultants, Phoenix, Arizona
  - Global Research Management, Glendale, California
  - Eye Research Foundation, Newport Beach, California